CLINICAL TRIAL: NCT00367666
Title: Evaluation of Multimodality Breast Imaging: Lesion Staging
Brief Title: Using Diagnostic Tools to Stage Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol 414500; NIH funded; NCT00194337 (obsolete NCT alias)
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography; Ultrasonography; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Diagnosed with Breast Cancer (Experimental)
  Interventions: Device: MRI, Digital Mammography, Ultrasound and Positron Emission Tomography (PET)

INTERVENTIONS:
Device: MRI, Digital Mammography, Ultrasound and Positron Emission Tomography (PET)

SUMMARY:
This project is aimed at investigating the relative diagnostic and synergy of four state of the art breast imaging techniques (magnetic resonance imaging (MRI), full-field digital mammography (DMAM), ultrasound, and positron emission tomography (PET)) with respect to determining the extent of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women recently diagnosed with Breast Cancer
* Will be undergoing surgery (after study) at the Hospital of the University of Pennsylvania

Exclusion Criteria:

* Contraindications to MRI
* previously diagnosed with breast cancer (in the smae breast) within the past 5 years
* Patients with known locally advanced cancer (prior to study entry) being treated with preoperative adjuvant therapy.
* Pregnant women

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-03-01 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-03-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Abass Alavi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States